CLINICAL TRIAL: NCT03163875
Title: Quality of Life,Anxity,Depression and Quality of Sleep in Patients With Chronic Urticaria
Brief Title: Quality of Life in Patients With Chronic Urticaria
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, AMAbdelgawad, principle investigator, Assiut University
Other Study IDs: ziad
Record Dates: First submitted 2017-05-15; First posted 2017-05-23 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Chronic Urticaria
Keywords: erythema; wheal formation; vascular reaction of the skin
MeSH Terms: conditions — Chronic Urticaria; Erythema | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Hospital Anxiety and Depression Scale — To assess the levels of depression and anxiety, quality of sleep and quality of life (QoL) in chronic urticaria patients, using an interdisciplinary approach combining interview/questionnaire-based psychiatric and dermatological evaluations

SUMMARY:
Urticaria is one of the most frequent presenting complaints in dermatology, allergy, and emergency departments. The term chronic urticaria (CU) is understood as the appearance of recurrent wheals more than twice a week for over 6 consecutive weeks .Urticaria is not a single disease but a reaction pattern that represents cutaneous mast cell degranulation, resulting in extravasation of plasma into the dermis. The incidence of chronic urticaria is unknown, but it is thought to occur in 0.1%-3% of the population

DETAILED DESCRIPTION:
Chronic urticaria signs and symptoms include: patches of red or white wheals, usually on the face, trunk, arms or legs. Wheals vary in size, change shape, and appear and fade repeatedly as the reaction runs its course. Itching is common, which may be severe. Swelling may occur that causes pain or burning (angioedema), especially inside the throat and around the eyes, cheeks, lips, hands, feet and genitals.

It is characterized by a tendency for signs and symptoms to flare with triggers such as heat, exercise and stress as well as a tendency for symptoms to recur frequently and unpredictably, sometimes for months or years The significance of chronic urticaria is sometimes trivialised because it is a non-life-threatening disease, but the condition can be very uncomfortable and interfere with sleep and daily activities. It is one of the most common and frustrating diseases for both patients and physicians Chronic urticaria has a major impact on quality of life (QoL) , with impact on activities of daily living. Chronic urticaria patients reportedly suffer considerable loss of energy, sleep disturbance and emotional upset as well as restrictions in the social life. Depression and anxiety are the most common psychiatric diagnoses. These psychiatric disorders could also influence QoL

ELIGIBILITY:
Inclusion Criteria:

Patients with chronic urticaria defined as a 6-week or longer history of daily or almost daily itchy cutaneous weals with individual lesions lasting less than 24 h.

Age between 18 and 60 years.

Exclusion Criteria:

Patients who are unable to understand the questions, are unwilling to complete the questionnaire, or who have a psychiatric disorder, or obstructive sleep apnea.

Patients with malignant or central nervous system disease. Patients with cognitive impairment due to a current cerebral or psychotic illness.

Patients with current psychotherapy . glucocorticoids therapy in the last month.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Antihistamines will be discontinued at least 72 h prior to evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2018-06-10 (Estimated); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
measure number of patients affected with depression and anxity | one year
  The levels of depression and anxiety will be assessed by Hospital Anxiety Depression Scale (HADS) .

IPD SHARING:
Plan to Share IPD: No